CLINICAL TRIAL: NCT04258150
Title: TRIPPLE-R: Phase 2 Study in Pretreated Patients With Advanced Pancreatic Cancer to Assess Efficacy of Ipilimumab, Nivolumab and Tocilizumab in Combination With Radiation
Brief Title: Ipilimumab, Nivolumab, Tocilizumab and Radiation in Pretreated Patients With Advanced Pancreatic Cancer
Acronym: TRIPPLE-R
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: primary endpoint was not met
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Inna Chen, MD, Principal investigator, Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GI 1950
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; nivolumab; Opdivo; ipilimumab; Yervoy; tocilizumab; RoACTEMRA; radiation; SBRT
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Nivolumab; Ipilimumab; tocilizumab

STUDY DESIGN:
Intervention Model Description: Initially, patients will be enrolled in the study to treatment with ipilimumab, nivolumab and tocilizumab in combination with SBRT, until 30 patients have been treated (Part A: Lead-in). This Part A: Lead-in involves Department of Oncology, Herlev and Gentofte Hospital, Copenhagen University Hospital, Denmark.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): SBRT of 15 Gy will be given on day 1 of the first cycle. Nivolumab 6 mg/kg (up to 480 mg maximum) will be given on day 1 (± 3 days) of each 14-day treatment cycle until the progression of disease or maximum of 48 weeks, discontinuation due to toxicity, withdrawal of consent. Ipilimumab 1 mg/kg will be given on day 1 (± 3 days) twice in total every 6 weeks. Nivolumab will be administered as an IV infusion over 60 (± 5) minutes and then, after a 30 minutes rest period, ipilimumab will be administered as an IV infusion over 30 (± 5) minutes. Tocilizumab 8 mg/kg is given IV on day 1 (± 3 days) over 1-hour, repeated every 4 weeks. Tocilizumab infusion over 30 minutes is allowed after 5. infusion in the absence of infusion related events.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: Tocilizumab; Radiation: SBRT

INTERVENTIONS:
Drug: Nivolumab — 6 mg/kg IV q4w
  Other Names: Opdivo®
Drug: Ipilimumab — 1 mg/kg IV twice q6w
  Other Names: Yervoy®
Drug: Tocilizumab — 8 mg/kg IV q4w
Radiation: SBRT — * A total dose of 15 Gy as a single fraction is prescribed as the mean dose to the PTV.
  * PTV should be covered by 95% isodose (PTV D99% > 95%).

SUMMARY:
Pancreatic cancer (PC) remains a dreadful disease due to its often advanced stage at diagnosis and poor sensitivity to chemotherapy. Progression after 1. line chemotherapy is inevitable in patients with advanced PC, and treatment options for patients who progress after 1. line chemotherapy are limited. Considering the emerging role of the tumor microenvironment (TME), the combination of checkpoint blocking antibodies with agents that target the inhibitory effects of the TME could lead to better responses in tumor historically resistant to checkpoint blocking antibody approaches. Inflammation is one of the hallmarks of cancer, and contributes to PC initiation, enhanced invasiveness and metastasis. The immune-modulating cytokine interleukin-6 (IL-6) facilitates the inflammation cascade and key pathways within the respective TME, among others promotion of tumor-induced immunosuppression and facilitation of metastasis. Thus, IL-6 inhibition approach can potentially directly affect the immunosuppressive TME compartment.

To explore the synergy of the proposed combinatorial approach, participants with locally advanced/metastatic pancreatic tumors who have progressed during or after at least 1 line of systemic chemotherapy in the metastatic setting will receive nivolumab and ipilimumab administered in combination with radiotherapy and tocilizumab. It is anticipated that this clinical study will inform the use of this 3-drug combination for further phase II and/or phase III clinical testing.

DETAILED DESCRIPTION:
This is a phase II study assessing ipilimumab, nivolumab and tocilizumab in combination with SBRT of 15 Gy in patients with locally advanced or metastatic PC whose disease has progressed on at least 1. line chemotherapy with either a 5-FU-containing and /or gemcitabine containing chemotherapy. The trial is designed as an investigator initiated prospective open-label study in patients with advanced PC to determine the efficacy and safety ipilimumab, nivolumab and tocilizumab in combination with SBRT.

This study will consist of Part A, Lead-in, as well as a possible Part B, non-randomized expansion (Part B: Expansion) or a possible Part B, randomized controlled study (Part B: RCT).

Initially, patients will be enrolled in the study to treatment with ipilimumab, nivolumab and tocilizumab in combination with SBRT, until 30 patients have been treated (Part A: Lead-in). Patient recruitment and tumor assessment will be monitored on an ongoing basis. This Part A: Lead-in involves Department of Oncology, Herlev and Gentofte Hospital, Copenhagen University Hospital, Denmark.

Multicenter extension will be activated in case of successfully completed lead-in phase and the format of that Part B will be determined based on the responses seen in the first 30 patients in Part A. A protocol amendment will be made if criteria are met to proceed to Part B. The protocol amendment will include available data from Part A and any changes to study design, additional sites and statistical plan, if needed.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent

  * Subjects must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care
  * Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study
* Histological or cytological confirmation of locally advanced or metastatic pancreatic carcinoma prior to entering this study
* Prior therapy requirements:

  * For Part A and Part B Expansion: there is no upper limit on the number of prior chemotherapy regimens received. Patients must have received and progressed during or after at least 1 line of systemic chemotherapy in the metastatic setting (gemcitabine or 5-FU based regimens).
  * For Part B RCT: patients must have tumor progression following prior standard first-line 5-FU-containing or gemcitabine-containing chemotherapy (no more than 1 prior chemotherapy regimen or any other systemic therapy for recurrent/metastatic pancreatic carcinoma).
  * Notes:

    * If a participant received adjuvant/neoadjuvant systemic combinational therapy, and progressed within 6 months, the adjuvant/neoadjuvant treatment will be considered as 1 line of systemic treatment.
    * In general, discontinuation of 1 drug in a multi-drug regimen and continuation of other drug(s), is considered part of the same line of treatment. Restarting the same regimen after a drug holiday or maintenance chemotherapy can also be considered part of the same line of treatment. Switching from IV (5-FU) to an oral formulation (capecitabine) of the same drug is also considered part of the same line of treatment
    * Minimum time from first systemic therapy for recurrent/metastatic adenocarcinoma of pancreas to progression should be at least 3 months
* Age 18 years and older
* ECOG/WHO Performance Status (PS) 0-1
* All participants will be required to undergo mandatory pre- and on-treatment biopsies at acceptable clinical risk as judged by the investigator. An archival pre-treatment sample is not acceptable.
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 10⁹/L
  * Platelet count ≥ 100 x 10⁹/L
  * Serum bilirubin ≤ 1.5 x upper limit of normal (ULN) (patients with Gilbert's Syndrome must have a total bilirubin ≤ 50 mmol/L)
  * AST/ALT ≤ 5 x ULN
  * Serum creatinine ≤ 1.5 x ULN or CrCl ≥ 40 mL/min (using the Cockcroft-Gault formula)
* Women of childbearing potential (WOCBP) must use method(s) of contraception as indicated in Appendix 3. For a teratogenic study drug and/or when there is insufficient information to assess teratogenicity (preclinical studies have not been done), a highly effective method(s) of contraception (failure rate of less than 1% per year) is required. The individual methods of contraception and duration should be determined in consultation with the investigator. WOCBP must follow instructions for birth control when the half-life of the investigational drug is greater than 24 hours, contraception should be continued for a period of 30 days plus the time required for the investigational drug to undergo five half-lives. The half-life of nivolumab and ipilimumab is up to 25 days and 18 days, respectively. WOCBP should therefore use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. The investigator shall review contraception methods and the time period that contraception must be followed. Men that are sexually active with WOCBP must follow instructions for birth control when the half-life of the investigational drug is greater than 24 hours, contraception should be continued for a period of 90 days plus the time required for the investigational drug to undergo five half-lives. The half-life of nivolumab is up to 25 days. Men who are sexually active with WOCBP must continue contraception for 31 weeks (90 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug. Women who are not of childbearing potential (i.e. who are postmenopausal or surgically sterile as well as azoospermic men do not require contraception
* Subjects must have signed and dated a BIOPAC approved written informed consent form in accordance with regulatory and institutional guidelines.

Exclusion Criteria:

* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results
* Participants with active, known or suspected autoimmune disease. Participants with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Current or prior use of immunosuppressive medication within 14 days before the first dose of ipilimumab, nivolumab and tocilizumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, or topical steroids; or local steroid injections (e.g. intra-articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g. CT scan premedication)
* Patients should be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Allergies and Adverse Drug Reaction

  * History of allergy to study drug components
  * History of severe hypersensitivity reaction to any monoclonal antibody
* WOCBP who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 12 months
  ORR in all patients using Investigator assessments according to RECIST 1.1

SECONDARY OUTCOMES:
Duration of response (DoR) | 12 months
  DoR in all patients using Investigator assessments according to RECIST 1.1.
Disease control rate (DCR) | 12 months
  DCR in all patients using Investigator assessments according to RECIST 1.1.
Progression free survival (PFS) | 12 months
  PFS in all patients using Investigator assessments according to RECIST 1.1.
Overall survival (OS) | 12 months
  OS in all patients using Investigator assessments according to RECIST 1.1.
EORTC QLQ-C30 | 12 months
  Adjusted mean change from baseline in global QoL score from the EORTC QLQ-C30 questionnaire.
Incidence of treatment-related AEs, SAEs, AEs leading to discontinuation, death, and laboratory abnormalities | 12 months
  AEs, physical examinations, laboratory findings (including clinical chemistry, hematology), vital signs (including blood pressure and pulse).

CONTACTS AND LOCATIONS:
Overall Officials: Inna M Chen, MD, Principal Investigator — Herlev Hospital
Locations (1):
- Herlev & Gentofte University Hospital, Denmark, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen IM, Donia M, Chamberlain CA, Jensen AWP, Draghi A, Theile S, Madsen K, Hasselby JP, Toxvaerd A, Hogdall E, Lorentzen T, Wilken EE, Geertsen P, Svane IM, Johansen JS, Nielsen D. Phase 2 study of ipilimumab, nivolumab, and tocilizumab combined with stereotactic body radiotherapy in patients with refractory pancreatic cancer (TRIPLE-R). Eur J Cancer. 2023 Feb;180:125-133. doi: 10.1016/j.ejca.2022.11.035. Epub 2022 Dec 10. PMID 36592507